CLINICAL TRIAL: NCT06475664
Title: Colorectal Cancer Legal and Administrative Burden Support: A Pilot Clinical Trial
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2023LS176
Record Dates: First submitted 2024-06-18; First posted 2024-06-26 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a single center single-arm, pilot study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): adult patients with advanced colorectal cancel
  Interventions: Other: Personalized legal care services

INTERVENTIONS:
Other: Personalized legal care services — Participants will receive free, personalized legal care services from Cancer Legal Care (CLC), a nonprofit organization located in the Twin Cities of Minnesota. The duration of study participation is 6 months, however, participants may continue to access free personalized legal care services beyond this period.

SUMMARY:
This is a single center single-arm, pilot study of proactive and early connection with free legal care services for persons with advanced colorectal cancer to assess the feasibility, acceptability, and preliminary efficacy of this intervention in improving financial and psychosocial outcomes. Participants will receive free, personalized legal care services from Cancer Legal Care (CLC), a nonprofit organization located in the Twin Cities of Minnesota. The duration of study participation is 6 months, however, participants may continue to access free personalized legal care services beyond this period. All participants continue to receive standard of care as prescribed by their treating physician.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of advanced stage colorectal cancer.
* Estimated life expectancy of over 6 months in the opinion of the treating oncologist.
* 18 years of age or older at the time of consent.
* Able to understand, speak, read, and write in English.
* Able to provide voluntary written consent prior to the performance of any research related activity.

Exclusion Criteria:

* Lacks capacity to consent/has diminished capacity to consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2024-10-18 (Actual); Study Completion 2025-06-05 (Actual)

PRIMARY OUTCOMES:
The Perceived Stress Scale 4 (PSS-4) | baseline, 3 months, 6 months
  A 4-item measure of perceived stress.
The Cancer Behavior Inventory-Brief Version (CBI-B) | baseline, 3 months, 6 months
  A 12-item measure of self-efficacy coping with cancer.
The COmprehensive Score for financial Toxicity (COST) | baseline, 3 months, 6 months
  A 12-item measure of financial toxicity.
The National Comprehensive Cancer Network's (NCCN) Distress Thermometer | baseline, 3 months, 6 months
  A single-item measure of psychological distress.
The Spitzer Uniscale (UNISCALE) | baseline, 3 months, 6 months
  A single-item measure of overall quality of life.
Patient Satisfaction with Interpersonal Relationship with Navigator (PSN-I) | baseline, 3 months, 6 months
  A 9-item measure of perceptions of interpersonal relationships with a patient navigator (i.e. CLC).
Pearlin Mastery Scale | baseline, 3 months, 6 months
  A 7-item measure of psychological coping
  (mastery).
The Life Engagement Test (LET) | baseline, 3 months, 6 months
  A 6-item measure of purpose in life, defined as the extent to which a person engages in activities that are personally meaningful.
Rosenberg Self-Esteem (RSE) Scale | baseline, 3 months, 6 months
  A 10-item measure of self-esteem.
Cancer Related Behavior Questionnaire | baseline, 3 months, 6 months
  A 31-item measure of comfort facing cancer related issues.
Cancer Legal Care Services Questionnaire | baseline, 3 months, 6 months
  A 13-item measure of CLC

CONTACTS AND LOCATIONS:
Overall Officials: Arjun Gupta, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States